CLINICAL TRIAL: NCT05516199
Title: Antenatal Breastmilk Expression From Week 34 of Gestation Safety in Pregnancy and Benefits for the Newborn Infant: A Pilot Randomized Study
Brief Title: Antenatal Breastmilk Expression From Week 34 of Gestation
Acronym: EXPRESS-MOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Marie Bendix Simonsen, M.D., Principal Investigator, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OUH-HCA005
Record Dates: First submitted 2022-08-11; First posted 2022-08-25 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Breastmilk Expression; Collection, Breastmilk; Breastfeeding; Healthy
Keywords: Infant nutrition; Lactation; Breastmilk; Breastfeeding
MeSH Terms: conditions — Breast Milk Expression; Breast Feeding

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antenatal breastmilk expression (Experimental): Breastfeeding consultation with trained midwife in week 33 + antenatal breastmilk expression from week 34
  Interventions: Behavioral: Antenatal breastmilk expression; Behavioral: Breastfeeding consultation
- Control (Other): Breastfeeding consultation with trained midwife in week 33
  Interventions: Behavioral: Breastfeeding consultation

INTERVENTIONS:
Behavioral: Antenatal breastmilk expression — Stimulation of the breast by hand/handexpression of breastmilk during pregnancy from week 34
  Arms: Antenatal breastmilk expression
Behavioral: Breastfeeding consultation — 60 min standardized breastfeeding consultation with a trained midwife, with focus on practical breastfeeding skills

SUMMARY:
In this pilot study, the investigators aim to examine if antenatal breastmilk expression from week 34 of pregnancy is a safe and feasible procedure for the mother and fetus. Furthermore, the investigators want to evaluate breastfeeding rates.

DETAILED DESCRIPTION:
In a randomized pilot study, 60 healthy pregnant women will be randomized either to antenatal breastmilk expression from week 34+0 until delivery or no antenatal breastmilk expression. Furthermore, all participants will have an individual breastfeeding consultation with a trained midwife in week 33 of pregnancy. At the consultation, the intervention group will also be taught how to perform antenatal expression by hand and store any expressed breastmilk correctly. All women included in this study will receive standard care.

To detect signs of uterine contractions or fetal reaction in relation to stimulation of the breast, a cardiotocography (CTG) will be performed before, during and after the first expression in the intervention group. If the CTG is normal the women can perform breastmilk expression by hand 5 minutes at each breast two times per day until birth, and collect and store any expressed milk.

During the intervention and 8 weeks after birth the participating women will receive weekly push-messages through an application on their smartphone. The messages include short questions about the handexpression of milk in pregnancy as well as regarding feeding of the infant after birth. At the end of the study the mothers will be invited for an interview to investigate their experience with the procedure, but this is an independent study and therefore not a part of this protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy nulliparous women with no major chronic or pregnancy related diseases
2. BMI <27
3. Danish speaking
4. Singleton pregnancies
5. Planning to exclusively breastfeed their infants and deliver at Odense University Hospital (Odense and Svendborg)

Exclusion Criteria:

1. Suspected fetal intrauterine growth restriction or known major fetal anomaly
2. Women at risk of preterm birth with one of the following diagnoses: Placenta previa, premature preterm rupture of membranes (PPROM) or previous cervical conization
3. Women taking medications where breastfeeding is contraindicated
4. Women with prior breast surgery: Breast reductive surgery or breast implants

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — No. They have to be able to be pregnant
Enrollment: 60 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Gestational age at birth in the two groups | Through study completion, an avarage of 1 year.
  Gestational age of infant at birth. Information will be found through medical records. In the weekly push-messages the women have to answer if they have been giving birth. If they click yes, investigators get a notification and find gestational age and baseline infant characteristics through medical records.

SECONDARY OUTCOMES:
Number of weekly breastmilk expressions before birth | Through study completion, an avarage of 1 year.
  Number of weekly expressions in interventiongroup. Measured through the weekly push-messages.
Amount of breastmilk expressed | Through out the study, an average of 1 year. Assesment when all women included have been giving birth.
  How many women will be capable of expressing any milk before birth in intervention group, and how many ml. Volume is measured by each women using a container with a mL scale and reported through weekly self reported push-messages.
Breastfeeding rates 1, 2, 4 and 8 weeks after birth | Through study completion, an avarage of 1 year.
  Measured through weekly self-reported push-messages in both groups
Number of exclusively breastfeeding versus partially breastfeeding women in each group at 1, 2, 4 and 8 weeks after birth | 1, 2, 4 and 8 weeks after birth
  Measured through the weekly self-reported push-messages in both groups
Adverse reactions from mother or fetus during first breastmilk expression | Through study completion, an avarage of 1 year.
  Contractions and/or fetal stimulation during the first breastmilk expression during pregnancy, assessed with CTG

CONTACTS AND LOCATIONS:
Overall Officials: Marie B Simonsen, M.D, Principal Investigator — OUH & SDU
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Time Frame: Study protocol, SAP and ICF after protocol publication. CSR: After ended intervention and data collection
Access Criteria: Write to principal investigator to request data. Data will be transferred to Rigsarkivet Denmark if possible with regard to GDP regulations.

REFERENCES:
- [Background] Ford SL, Lohmann P, Preidis GA, Gordon PS, O'Donnell A, Hagan J, Venkatachalam A, Balderas M, Luna RA, Hair AB. Improved feeding tolerance and growth are linked to increased gut microbial community diversity in very-low-birth-weight infants fed mother's own milk compared with donor breast milk. Am J Clin Nutr. 2019 Apr 1;109(4):1088-1097. doi: 10.1093/ajcn/nqz006. PMID 30982856
- [Background] Wagner KJP, Rossi CE, Hinnig PF, Alves MA, Retondario A, Vasconcelos FAG. ASSOCIATION BETWEEN BREASTFEEDING AND OVERWEIGHT/OBESITY IN SCHOOLCHILDREN AGED 7-14 YEARS. Rev Paul Pediatr. 2021 Feb 24;39:e2020076. doi: 10.1590/1984-0462/2021/39/2020076. eCollection 2021. PMID 33656144
- [Background] Laine MK, Kautiainen H, Gissler M, Pennanen P, Eriksson JG. Impact of gestational diabetes mellitus on the duration of breastfeeding in primiparous women: an observational cohort study. Int Breastfeed J. 2021 Feb 16;16(1):19. doi: 10.1186/s13006-021-00369-1. PMID 33593367
- [Background] Victora CG, Bahl R, Barros AJ, Franca GV, Horton S, Krasevec J, Murch S, Sankar MJ, Walker N, Rollins NC; Lancet Breastfeeding Series Group. Breastfeeding in the 21st century: epidemiology, mechanisms, and lifelong effect. Lancet. 2016 Jan 30;387(10017):475-90. doi: 10.1016/S0140-6736(15)01024-7. PMID 26869575
- [Background] Ballard O, Morrow AL. Human milk composition: nutrients and bioactive factors. Pediatr Clin North Am. 2013 Feb;60(1):49-74. doi: 10.1016/j.pcl.2012.10.002. PMID 23178060
- [Background] Yu X, Li J, Lin X, Luan D. Association between Delayed Lactogenesis Ⅱ and Early Milk Volume among Mothers of Preterm Infants. Asian Nurs Res (Korean Soc Nurs Sci). 2019 May;13(2):93-98. doi: 10.1016/j.anr.2019.02.001. Epub 2019 Feb 16. PMID 30776448
- [Background] Underwood MA. Human milk for the premature infant. Pediatr Clin North Am. 2013 Feb;60(1):189-207. doi: 10.1016/j.pcl.2012.09.008. Epub 2012 Oct 18. PMID 23178065
- [Background] Parker LA, Sullivan S, Krueger C, Mueller M. Association of timing of initiation of breastmilk expression on milk volume and timing of lactogenesis stage II among mothers of very low-birth-weight infants. Breastfeed Med. 2015 Mar;10(2):84-91. doi: 10.1089/bfm.2014.0089. Epub 2015 Feb 6. PMID 25659030
- [Background] Forster DA, Moorhead AM, Jacobs SE, Davis PG, Walker SP, McEgan KM, Opie GF, Donath SM, Gold L, McNamara C, Aylward A, East C, Ford R, Amir LH. Advising women with diabetes in pregnancy to express breastmilk in late pregnancy (Diabetes and Antenatal Milk Expressing [DAME]): a multicentre, unblinded, randomised controlled trial. Lancet. 2017 Jun 3;389(10085):2204-2213. doi: 10.1016/S0140-6736(17)31373-9. PMID 28589894
- [Background] Lopez-Fernandez G, Barrios M, Goberna-Tricas J, Gomez-Benito J. Breastfeeding during pregnancy: A systematic review. Women Birth. 2017 Dec;30(6):e292-e300. doi: 10.1016/j.wombi.2017.05.008. Epub 2017 Jun 19. PMID 28642112
- [Background] Lamba S, Chopra S, Negi M. Effect of Antenatal Breast Milk Expression at Term Pregnancy to Improve Post Natal Lactational Performance. J Obstet Gynaecol India. 2016 Feb;66(1):30-4. doi: 10.1007/s13224-014-0648-7. Epub 2015 Jan 20. PMID 26924904
- [Background] Foudil-Bey I, Murphy MSQ, Dunn S, Keely EJ, El-Chaar D. Evaluating antenatal breastmilk expression outcomes: a scoping review. Int Breastfeed J. 2021 Mar 12;16(1):25. doi: 10.1186/s13006-021-00371-7. PMID 33712049
- [Background] Casey JRR, Banks J, Braniff K, Buettner P, Heal C. The effects of expressing antenatal colostrum in women with diabetes in pregnancy: A retrospective cohort study. Aust N Z J Obstet Gynaecol. 2019 Dec;59(6):811-818. doi: 10.1111/ajo.12966. Epub 2019 Mar 19. PMID 30891743
- [Background] Demirci JR, Glasser M, Fichner J, Caplan E, Himes KP. "It gave me so much confidence": First-time U.S. mothers' experiences with antenatal milk expression. Matern Child Nutr. 2019 Oct;15(4):e12824. doi: 10.1111/mcn.12824. Epub 2019 May 23. PMID 30950165
- [Background] Demirci J, Schmella M, Glasser M, Bodnar L, Himes KP. Delayed Lactogenesis II and potential utility of antenatal milk expression in women developing late-onset preeclampsia: a case series. BMC Pregnancy Childbirth. 2018 Mar 15;18(1):68. doi: 10.1186/s12884-018-1693-5. PMID 29544467
- [Background] Soltani H, Scott AM. Antenatal breast expression in women with diabetes: outcomes from a retrospective cohort study. Int Breastfeed J. 2012 Dec 1;7(1):18. doi: 10.1186/1746-4358-7-18. PMID 23199299
- [Result] Bruun S, Wedderkopp N, Molgaard C, Kyhl HB, Zachariassen G, Husby S. Using text messaging to obtain weekly data on infant feeding in a Danish birth cohort resulted in high participation rates. Acta Paediatr. 2016 Jun;105(6):648-54. doi: 10.1111/apa.13382. Epub 2016 Apr 13. PMID 26928297
- [Derived] Simonsen MB, Bentzen SB, Moller S, Holm KG, Vinter CA, Zachariassen G. Safety of antenatal breastmilk expression from week 34 of pregnancy: a randomized controlled pilot study (The Express-MOM study). Matern Health Neonatol Perinatol. 2025 Jan 3;11(1):2. doi: 10.1186/s40748-024-00197-1. PMID 39748396
- [Derived] Bentzen SB, Simonsen MB, Zachariassen G, Vinter CA, Garne Holm K. Women's bodily experience of antenatal breastmilk expression from 34 weeks of gestation: Qualitative results from the Express-MOM study. Eur J Midwifery. 2024 Nov 1;8. doi: 10.18332/ejm/193601. eCollection 2024. PMID 39493541

DOCUMENTS (2):
  • Study Protocol (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT05516199/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT05516199/SAP_001.pdf